CLINICAL TRIAL: NCT02121418
Title: Decitabine Plus Cytarabine for Induction of Remission in Newly Diagnosed Elderly Acute Myeloid Leukemia (AML) and Advanced Myelodysplastic Syndrome (MDS)
Brief Title: Decitabine and Cytarabine in Treating Older Patients With Newly Diagnosed Acute Myeloid Leukemia, High Risk Myelodysplastic Syndrome, or Myeloproliferative Neoplasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9019; NCI-2014-00769 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9019 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Chronic Myelomonocytic Leukemia-2; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders | interventions — Cytarabine; Decitabine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (decitabine, cytarabine) (Experimental): Patients receive decitabine IV daily on days 1-10 and cytarabine IV QD on days 1-7. Treatment repeats every 28-35 days for 2 courses in the absence of disease progression or unacceptable toxicity. After course 3, patients achieving remission will receive 1-2 more courses of therapy at the same dose. Patients in remission with significant side effects will receive decitabine and cytarabine at decreased doses. Patients not achieving remission will not receive any more treatment.
  Interventions: Drug: Cytarabine; Drug: Decitabine; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies decitabine and cytarabine in treating older patients with newly diagnosed acute myeloid leukemia, myelodysplastic syndrome that is likely to come back or spread to other places in the body, or myeloproliferative neoplasm. Drugs used in chemotherapy, such as decitabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving decitabine and cytarabine may work better than standard therapies in treating cancers of the bone marrow and blood cells, such as acute myeloid leukemia, myelodysplastic syndrome, or myeloproliferative neoplasm.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Examine whether a combination of decitabine given for 10 days (days 1-10), rather than the usual 5 days, plus "standard dose cytarabine (ara-C) (100 mg/m^2 daily days 1-7) might improve 6-month survival probability from the historical 65% to 80% in patients age >= 60 with newly diagnosed acute myeloid leukemia (AML).

II. Test whether this combination might maintain complete response (CR) rate at our historic 45% in these patients.

III. Study factors that lead physicians to escalate or maintain ara-C doses in those patients who have had an "intermediate response" short of CR to the first 2 cycles of the combination.

IV. While maintaining awareness of confounding covariates, examine the effect of such dose escalation on CR rate.

OUTLINE:

Patients receive decitabine intravenously (IV) daily on days 1-10 and cytarabine IV once daily (QD) on days 1-7. Treatment repeats every 28-35 days for 2 courses in the absence of disease progression or unacceptable toxicity. After course 3, patients achieving remission will receive 1-2 more courses of therapy at the same dose. Patients in remission with significant side effects will receive decitabine and cytarabine at decreased doses. Patients not achieving remission will not receive any more treatment.

After completion of study treatment, patients are followed up for 6 months and then periodically.

ELIGIBILITY:
Inclusion Criteria:

* Newly-diagnosed AML by World Health Organization (WHO) criteria (>= 20% myeloid blasts by morphology in either blood or marrow)
* High-risk myelodysplastic syndrome (MDS) or myeloproliferative neoplasm (MPN) including chronic myelomonocytic leukemia 2 (CMML2) as defined by 10-19% myeloid blasts in either blood or marrow
* Patients may have received azacitidine, decitabine, or lenalidomide but no "cytotoxic therapy" such as ara-C or anthracyclines; data suggest that failure to respond to azacitidine reduces probability of response to 3+7; hence in the interest of having a relatively homogeneous population, while patients who have received and failed azacitidine or decitabine will be eligible for this study, they will be analyzed separately from patients who have not received these drugs
* Treatment related mortality (TRM) score < 22.9; patients with TRM scores > 13.1, in whom the risk of death within 28 days of beginning induction therapy has averaged 41%, will preferentially be placed on protocol 2642
* Provision of written informed consent
* Note, unlike pharmaceutical company sponsored protocols eligibility is not conditioned on bilirubin, creatinine, or absence of other malignancy within the past 2-3 years; the TRM score incorporates creatinine and thus a high creatinine can in principle be offset by favorable values for the other covariates in the TRM score; bilirubin was not a covariate in the TRM; furthermore, in the doses we are using, dose adjustment of decitabine or ara-C is not indicated in the presence of renal or hepatic abnormalities; our broad eligibility criteria may increase the likelihood that our results will be generalizable; the inability to reproduce results of early phase AML studies has been a problem in the past

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2017-02-08 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (9):
- United States (9):
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Group Health Cooperative, Redmond, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Decitabine, Cytarabine): Patients receive decitabine IV daily on days 1-10 and cytarabine IV QD on days 1-7. Treatment repeats every 28-35 days for 2 courses in the absence of disease progression or unacceptable toxicity. After course 3, patients achieving remission will receive 1-2 more courses of therapy at the same dose. Patients in remission with significant side effects will receive decitabine and cytarabine at decreased doses. Patients not achieving remission will not receive any more treatment. 12 patients were consented and treated.
Period: Overall Study
Arm/Group | Treatment (Decitabine, Cytarabine)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Decitabine, Cytarabine)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival of Patients Over Age 60 With Newly Diagnosed AML/High Risk MDS
Description: Compared to historical data of a completed Southwestern Oncology Group (SWOG) trial of azacitidine and gemtuzumab ozogamicin.
Time Frame: At 6 months
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine, Cytarabine)
Number analyzed (Participants) | 12
participants | 7

2. Secondary Outcome: Response Rate
Description: Rate of Complete Response or Complete Response with Incomplete Count Recovery
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (Decitabine, Cytarabine)
Number analyzed (Participants) | 12
participants
  Complete Respnose | 4
  Complete Response with Incomplete Count Recovery | 3

ADVERSE EVENTS:
Time Frame: 2 years
Description: Other [not including serious] adverse events were not addressed.
Arm/Group | Treatment (Decitabine, Cytarabine)
All-Cause Mortality (participants affected / at risk) | 9/12
Serious Adverse Events (participants affected / at risk) | 11/12
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Decitabine, Cytarabine) (N=12)
Febrile Neutropenia (Infections and infestations) | 4 (5)
Pneumonia (Infections and infestations) | 6 (6)
MRSA Bacteremia (Infections and infestations) | 1 (1)
Hyponatremia (Investigations) | 1 (1)
Hypertension (Blood and lymphatic system disorders) | 1 (1)
Staph Bacteremia (Infections and infestations) | 2 (2)
Hypokalemia (Investigations) | 1 (1)
Right cheek cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Bacterial Liver Abscess (Hepatobiliary disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Syncope (Cardiac disorders) | 1 (1)
C. Difficile Diarrhea (Infections and infestations) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyomyositis of B/L calf (Infections and infestations) | 1 (1)
Afibrillation (Cardiac disorders) | 1 (1)
Hypoxia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hyperbilirubinemia (Investigations) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Esophagogastric mucosal junction ulcer (Gastrointestinal disorders) | 1 (1)
Clostridium Ramosum bacteremia (Infections and infestations) | 1 (1)
Rothia Bacteremia (Infections and infestations) | 1 (1)
Oral mucositis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT02121418/Prot_SAP_000.pdf